CLINICAL TRIAL: NCT03232788
Title: Use of Computer Aided Design-Computer Aided Manufacturing and Additively Manufactured Scaffolds for Treatment of Gingival Recession Associated With Interproximal Tissue Deficiency
Brief Title: Use of Scaffolds for Treatment of Gingival Recession Associated With Interproximal Tissue Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vitor de Toledo Stuani, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOB3DPrint1
Record Dates: First submitted 2017-07-23; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Recession; Periodontal Diseases
Keywords: Periodontal disease; Recession; Black space
MeSH Terms: conditions — Periodontal Diseases | interventions — Bone Regeneration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Bone regeneration with autogenous bone + scaffold.
  Interventions: Procedure: Bone regeneration; Device: Scaffold
- Control group (Active Comparator): Bone regeneration with autogenous bone + collagen membrane.
  Interventions: Procedure: Bone regeneration; Device: Collagen membrane

INTERVENTIONS:
Procedure: Bone regeneration — Autogenous bone will be placed over periodontal defect after root treatment with scaling and root planing.
Device: Collagen membrane — A collagen membrane will be used to cover the autogenous bone.
  Arms: Control group
Device: Scaffold — A hydroxyapatite and polycaprolactone scaffolds will be used to cover the autogenous bone.
  Arms: Test group

SUMMARY:
This study will seek to evaluate the predictability and efficacy of a Computer Aided Design-Computer Aided Manufacturing and additively manufactured polycaprolactone and hydroxyapatite scaffolds in these defects compared to traditional guided tissue regeneration. 40 gingival recessions associated with interproximal tissue deficiency will be divided into two groups: control group (autogenous bone + collagen membrane; n = 20) and test group (autogenous bone + scaffold; n = 20).

DETAILED DESCRIPTION:
The treatment of gingival recessions associated with interproximal bone and gingival tissue deficiency, and also the absence of interdental papilla, are major challenges within the periodontics due to lacking predictability. However, an intervention in these cases is extremely important, since the presence of these defects is associated with aesthetic, phonetic, hypersensitivity and may be associated with other dental damages. This study will seek to evaluate the predictability and efficacy of a Computer Aided Design-Computer Aided Manufacturing and additively manufactured polycaprolactone and hydroxyapatite scaffolds in these defects compared to traditional guided tissue regeneration. 40 gingival recessions associated with interproximal tissue deficiency will be divided into two groups: control group (autogenous bone + collagen membrane; n = 20) and test group (autogenous bone + scaffold; n = 20). A split-mouth design will be used with both procedures performed at the same surgical time.

ELIGIBILITY:
Inclusion Criteria:

* Presenting at least two single-rooted teeth with Miller's Class III and IV recessions with Norland & Tarnow class I, II or III papilla deficiency

Exclusion Criteria:

* History of periodontal surgery at the area on the last 12 months
* Use of drugs that affect periodontal tissues (eg: anticonvulsants, calcium channel blockers, cyclosporine, bisphosphonates, hormone-based contraceptives, steroids)
* Pregnant
* Smokers
* Diabetics
* History of head and neck radiotherapy
* Teeth without adjacent mesial and distal contact
* Teeth with mobility
* Malpositioned teeth
* Teeth with endodontic treatment
* Teeth without a visible cementoenamel junction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Total root coverage measured with a periodontal probe in millimeters | One year
  Ideal if the distance from cemento-enamel junction to gingival margin = 0 mm
Total interdental papilla formation measured with a periodontal probe in mm | One year
  Ideal if the distance from dental contact point to interdental papilla top = 0 mm

SECONDARY OUTCOMES:
Depth of probing measured with a periodontal probe in millimeters | One year
  The distance from gingival margin and the apical point of gingival pocket or sulcus
Clinical attachment level measured with a periodontal probe in millimeters | One year
  The distance from cemento-enamel junction and the apical point of gingival pocket or sulcus
Gingival bleeding index measured with a periodontal probe | One year
  Evaluated by the presence or absence of bleeding after probing
Radiographic bone formation measured digitally in millimeters | One year
  The distance from interdental bone crest and cemento-enamel junction
Tomographic bone formation measured digitally in cubic millimeters | One year
  The variation of bone volume observed by tomography digital reconstruction
Evaluation of pink aesthetics by professionals using the Pink Esthetic Score | One year
  Photographic evaluation of gingival aesthetics during the treatment done by blinded periodontists.
Patient's evaluation of aesthetics using a visual analogue scale | One year
  Patient's aesthetic evaluation with a score ranging from 0 (terrible aesthetic) to 10 (excellent aesthetic)
Patient's evaluation of dental sensibility using a visual analogue scale | One year
  Patient's dental sensibility evaluation with a score ranging from 0 (no sensibility) to 10 (intense sensibility)
Patient's evaluation of post-operatory pain using a visual analogue scale | 1 month
  Patient's post-operatory pain evaluation with a score ranging from 0 (no pain) to 10 (intense pain)

CONTACTS AND LOCATIONS:
Overall Officials: Vitor T Stuni, MSc, Principal Investigator — PhD student
Locations (1):
- Bauru School of Dentistry - University of Sao Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided